CLINICAL TRIAL: NCT06765460
Title: Effectiveness of Medical Prescription of Exercise in Children to Increase Physical Activity Levels.
Brief Title: Prescription of Exercise in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Virgen de las Nieves (Other)
Responsible Party: Principal Investigator, Ángel Morillas Mingorance, Médico pediatra, University Hospital Virgen de las Nieves
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Zaidin exercises
Record Dates: First submitted 2024-12-23; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-12

CONDITIONS: Children; Exercise; Physical Activity; Screen Time
Keywords: children; exercise; physical activity; Screen time
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: A randomized controlled clinical trial with parallel groups was conducted, including 130 participants aged 6 to 14 years. Data on PA levels (duration and intensity), ST, and anthropometric measures were collected via questionnaire. Participants were divided into two groups: HA (3 minutes) and medical prescription of exercise [MPE] (10 minutes). PA levels were assessed at 3 and 12 months, with results recorded using the same questionnaire. A multivariate data analysis was performed
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: restrictive block randomization conducted using STATA version 16 software. Those within the intervention group received an individualized MPE, while participants in the control group received brief HA. To avoid classification bias in terms of PA level measurement, both the randomly selected intervention (HA and MPE) and the subsequent data collection (baseline, at 3 months and 12 months) were performed by the same blinded investigator, ensuring data consistency and validity. Participants did not know which intervention they were receiving as they did not know the actual recomendations in pediatric patients about exercise and screen time
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Medical prescription of exercise (MPE) (Experimental): MPE consists of dedicating a specific time to establish a specific and individualized exercise plan for the patient, with the premises of fully assessing their physical fitness, motivation, adaptability to change and the possibility of exercising within their social environment, as well as the achievement of specific objectives within an agreed follow-up period.
  Interventions: Behavioral: Medical prescription of exercise
- Health Advice (HA) (Active Comparator): providing the patient with information and motivation in line with general international recommendations to try to increase PA levels in their daily life. This advice can be given in a short period of time (up to three minutes) during any medical consultation
  Interventions: Behavioral: Health Advice

INTERVENTIONS:
Behavioral: Medical prescription of exercise — MPE consists of dedicating a specific time to establish a specific and individualized exercise plan for the patient, with the premises of fully assessing their physical fitness, motivation, adaptability to change and the possibility of exercising within their social environment, as well as the achievement of specific objectives within an agreed follow-up period
  Arms: Medical prescription of exercise (MPE)
Behavioral: Health Advice — HA consists of providing the patient with information and motivation in line with general international recommendations to try to increase PA levels in their daily life. This advice can be given in a short period of time (up to three minutes) during any medical consultation
  Arms: Health Advice (HA)

SUMMARY:
Most pediatric populations do not meet the physical activity (PA) recommendations set by international organizations. The effectiveness of casual PA advice provided during medical consultations has not been adequately assessed for its role in fostering this healthy habit. This study aims to evaluate the effectiveness of medical prescriptions for PA in increasing PA levels in children compared to standard health advice (HA), as well as measuring the effectiveness of these recommendations in reducing daily screen time (ST) in the pediatric population. A randomized controlled clinical trial with parallel groups was conducted, including 130 participants aged 6 to 14 years. Data on PA levels (duration and intensity), ST, and anthropometric measures were collected via questionnaire. Participants were divided into two groups: HA (3 minutes) and medical prescription of exercise [MPE] (10 minutes). PA levels were assessed at 3 and 12 months, with results recorded using the same questionnaire. A multivariate data analysis was performed. Further research is needed to develop effective and sustainable public health interventions to prevent long-term sedentary behavior in children.

DETAILED DESCRIPTION:
* Both HA and MPE interventions could effectively increase children's PA duration and intensity, resulting in a higher PA classification range.
* An inverse relationship may be identified between ST and PA, suggesting that reducing ST could encourage healthier habits in children.
* Pediatricians play a pivotal role in promoting lifestyle changes through brief yet targeted interventions, significantly influencing children's PA levels and reducing ST. These findings highlight the need for further research to optimize public health initiatives within pediatric care.

ELIGIBILITY:
Inclusion Criteria:

We included pediatric patients between 6 and 14 years of age who were part of two pediatric PC groups of an urban health centre in Granada (Spain) who attended a face-to-face consultation of any type.

Exclusion Criteria:

chronic or complex pathology preventing moderate or intense physical activity or those who did not give consent

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 130 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Efectiveness of MPE and HA | from enrollment to 12 months
  test whether brief HA and/or individualized MPE in PC increases physical activity levels in childhood.

CONTACTS AND LOCATIONS:
Locations (1):
- Avenida de las Fuerzas Armadas, 2, 18014, Granada, Granada, Granada, Spain

IPD SHARING:
Plan to Share IPD: Yes
Permission to reproduce material from other sources: Specific permissions and related documentation are available upon request
Supporting Information: Study Protocol, SAP, ICF